CLINICAL TRIAL: NCT01281956
Title: A Phase II Clinical Trial of PRX-00023 Therapy in Localization-Related Epilepsy
Brief Title: PRX-00023 Therapy in Localization-Related Epilepsy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 110039; 11-N-0039
Record Dates: First submitted 2011-01-21; First posted 2011-01-24 (Estimated); Results first posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2017-10-05

CONDITIONS: Epilepsy; Epilepsy, Temporal Lobe; Partial Epilepsy
Keywords: Epilepsy; Drug Trial; Serotonin; Serotonin 1A Receptor; Temporal Lobe Epilepsy; Partial Epilepsy
MeSH Terms: conditions — Epilepsy; Epilepsy, Temporal Lobe; Epilepsies, Partial | interventions — naluzotan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo Then PRX (Experimental): Subjects are administered Placebo x3 months followed by PRX (selective 5HT1A agonist) x3 months
  Interventions: Drug: PRX-00023; Drug: Placebo
- PRX Then Placebo (Experimental): Subjects are administered PRX (selective 5HT1A agonist) x3 months followed by Placebo x3 months
  Interventions: Drug: PRX-00023; Drug: Placebo

INTERVENTIONS:
Drug: PRX-00023 — PRX-00023 (Selective 5HT1A agonist)
Drug: Placebo — Placebo

SUMMARY:
Background:

- The brain chemical serotonin helps nerve cells communicate. Previous research suggests that serotonin activity may be lower in brain areas where seizures start, and that increasing activity at the serotonin receptor site on nerve cells may help prevent seizures. Researchers are interested in determining whether the experimental medication PRX-00023, which increases the activity of serotonin receptors, can reduce seizure frequency in people whose seizures are not well-controlled on antiseizure medication. PRX-00023 has not previously been studied in people with epilepsy and has not previously been given to people taking antiseizure medication at the same time.

Objectives:

- To evaluate the effectiveness of PRX-00023 in reducing the frequency of epileptic seizures that start from only one part of the brain.

Eligibility:

- Individuals between 18 and 65 years of age who have frequent epileptic seizures even after trying at least two different standard anti-seizure medications (either at the same time or one after the other).

Design:

* The study requires 9 outpatient visits to the NIH Clinical Center over a 34-week period. Individuals who choose to participate in additional studies may be an inpatient during some of these visits.
* Participants will be screened with a medical history and physical examination, blood and urine samples, ECG, EEG, neuropsychological studies, imaging studies, including PET and MRI scans
* Participants will have a 6-week observation and evaluation period before starting the study medication. Participants who have at least four seizures during this period will be eligible for the treatment portion of the study.
* All participants will receive either PRX-00023 or a placebo pill twice daily for 12 weeks, and will have regular clinic visits with blood samples and imaging studies.
* After the 12-week period, participants will have a 2- to 3-week washout period without any study medication.
* Participants will then have another study medication period, and will receive the opposite pill (PRX-00023 or placebo) from the one taken in the first treatment phase. Participants will continue to have regular clinic visits with blood samples, ECG, EEG and neuropsychologicalstudies.
* One month after the end of the second study medication phase, participants will have a followup evaluation with a physical examination, blood tests, ECG, EEG, mood and neuropsychological tests.

Outcome measures:

The primary outcome measure for drug efficacy will be:

Mean difference in seizure frequency comparing the active and placebo periods.

Secondary outcome measures for efficacy will be:

Proportion of patients with greater than or equal to 50% lower seizure rate on PRX-00023 than placebo

Hamilton Depression and Anxiety Rating scales

Performance on mood and neuropsychological testing scales

DETAILED DESCRIPTION:
Introduction:

PRX-00023 is a selective 5HT1A agonist being developed as an oral therapeutic treatment for epilepsy.

Objective:

To initiate a pilot clinical trial assessing the safety, tolerability and efficacy of the 5HT1A receptor agonist PRX-00023 in patients with localization-related epilepsy. PRX-00023 is a 5HT1A receptor agonist that has shown promise in clinical trials of depression. Patients with localization-related epilepsy have reduced 5HT1A receptor binding on 18FCWAY positron emission tomography (PET). Increasing neurotransmitter activity at 5HT1A receptor sites might ameliorate seizures. Moreover, depression is a common co-morbidity in people with epilepsy. Altered 5HT1A receptor binding has been found in depression.

Study Population:

Thirty adults with localization-related epilepsy.

Design:

A randomized, double-blind, placebo-controlled cross-over, phase II clinical trial. Subjects will be screened under protocol 01-N-0139 and will undergo medical and epilepsy history and physical examination, vital signs, ECG, clinical laboratory studies including standard clinical chemistry and hematology studies, urinalysis, pregnancy test for females of childbearing potential, and MRI scan and eo EEG monitoring will be performed if not previously completed successfully, and measurement of plasma AED levels (for those AEDs in which an assay is available at NIH).

The trial will have a baseline phase, which will last up to 6 weeks. Baseline may occur concurrent with screening procedures. The baseline phase will include measurement of seizure frequency (patient will record via seizure calendar). In addition the following will be administered, unless previously completed: Columbia Suicide Severity Rating Scale, neuropsychological and mood evaluations, FCWAY PET (if not already performed), EEG, measurement of plasma AED levels (if assay available), and pregnancy test (for women of child bearing potential), saliva samples will be obtained for genetic testing (if not previously obtained) and blood samples will be obtained during the PET procedure for cortisol and ACTH levels.

Following baseline, patients will begin the treatment phase (consisting of Period 1 and Period 2). Patients will be randomized to PRX-00023 (120mg BID) or matching placebo. After completion of the first treatment period, patients will undergo a washout period after which patients will be crossed over to the alternate treatment period.

Outcome measures:

1. Seizure frequency counts during the 3-month placebo and active treatment phases
2. Neuropsychological and mood indices
3. Safety assessment will include adverse events, vital signs, laboratory signs and physical examination.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Enrolled in protocol 01-N-0139
  2. Age 18 to 65
  3. Localization-related epilepsy diagnosed by standard clinical criteria that has not responded to treatment with up to two standard antiepileptic drugs either sequentially or in combination.
  4. Patients must be able to provide informed consent.
  5. Patients must be able to remain on their baseline AED drugs and doses for the duration of the study
  6. Patients must be able to use seizure calendars to record seizures throughout the trial.
  7. Experiences 4 seizures within a 6-week period

EXCLUSION CRITERIA:

1. Pregnancy or lactation
2. Women of child-bearing potential and men who are unable or unwilling to take adequate contraceptive precautions, including one of the following:

   * hormonal contraception (birth control pills, injected hormones or vaginal ring);
   * intrauterine device;
   * barrier methods (condom or diaphragm) combined with spermicide;
   * surgical sterilization (hysterectomy, tubal ligation, or vasectomy in a partner
3. Current treatment for another significant medical disorder, such as diabetes, or heart disease, or an untreated disorder, that is discovered during the screening examination and might interfere with the study and is determined by the PI to warrant exclusion of the participant.
4. An abnormality on clinical laboratory tests, physical examination, EEG or ECG that might increase the risk associated with trial participation or investigational product administration, such as hepatic enzyme elevation greater than twice normal, or hematocrit lower than 30.
5. A level 4 or 5 on the Columbia Suicide Severity Rating Scale rating for symptoms during the last month
6. Concomitant treatment with more than 2 AEDs
7. Evidence for a potentially progressive neurologic disorder, such as an astrocytoma
8. Use of sublingual lorazepam for seizure clusters more than once per wee
9. Use of any of the following prohibited medications/classes with less than required interval period:

   * Any other Investigational drugs; required interval period (weeks prior to baseline) is 4
   * benzodiazepines; required interval period (weeks prior to baseline) is 4
   * MAO Inhibitors anti depressant; required interval period (weeks prior to baseline) is 4
   * Buspirone; required interval period (weeks prior to baseline) is 2
   * other psychotropic medicines; required interval period (weeks prior to baseline) is 2
   * potent CYP3A4 inducers/inhibitors; required interval period (weeks prior to baseline) is 2 for:

     * Itraconazole
     * ketoconazole
     * HIV antivirals
     * clarithromycin
     * phenytoin
   * Prornolol is 2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-01-07; Primary Completion 2017-10-05 (Actual); Study Completion 2017-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William H Theodore, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Clinckers R, Smolders I, Meurs A, Ebinger G, Michotte Y. Anticonvulsant action of hippocampal dopamine and serotonin is independently mediated by D and 5-HT receptors. J Neurochem. 2004 May;89(4):834-43. doi: 10.1111/j.1471-4159.2004.02355.x. PMID 15140183
- [Background] Giovacchini G, Toczek MT, Bonwetsch R, Bagic A, Lang L, Fraser C, Reeves-Tyer P, Herscovitch P, Eckelman WC, Carson RE, Theodore WH. 5-HT 1A receptors are reduced in temporal lobe epilepsy after partial-volume correction. J Nucl Med. 2005 Jul;46(7):1128-35. PMID 16000281
- [Background] Hasler G, Bonwetsch R, Giovacchini G, Toczek MT, Bagic A, Luckenbaugh DA, Drevets WC, Theodore WH. 5-HT1A receptor binding in temporal lobe epilepsy patients with and without major depression. Biol Psychiatry. 2007 Dec 1;62(11):1258-64. doi: 10.1016/j.biopsych.2007.02.015. Epub 2007 Jun 22. PMID 17588547

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants that were consented to the protocol, did not participate in the study procedures. One participant was screened but was not randomized and did not receive study drug or placebo and one participant did not return for screening visit.
Groups:
- Placebo Then PRX: Participants with epilepsy receiving placebo during the first period followed by PRX during the second period
- PRX Then Placebo: Participants with epilepsy receiving PRX during the first period followed by Placebo during the second period
Period: 1st Intervention (3 Months)
Arm/Group | Placebo Then PRX | PRX Then Placebo
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: 2nd Intervention (3 Months)
Arm/Group | Placebo Then PRX | PRX Then Placebo
Started | 5 | 5
Completed | 4 | 5
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants Enrolled in Study: All participants enrolled in the study
Arm/Group | All Participants Enrolled in Study
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (12.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Seizure Frequency in the Active and Placebo Periods
Description: Participants used a seizure calendar to record the number of seizures that occurred during the three month treatment period, i.e., while participants were either on PRX-0023 or Placebo. Seizure frequency was calculated as the total number of seizures occurring during each three month period. For each period a mean was calculated across subjects.
Time Frame: Three months
Measure: Mean (Standard Deviation); unit: number of seizures
Groups:
- PRX-0023: Participants with epilepsy receiving PRX-0023
- Placebo: Participants with epilepsy receiving Placebo
Arm/Group | PRX-0023 | Placebo
Number analyzed (Participants) | 9 | 10
number of seizures | 66.6 (93.3) | 54.3 (79.7)

2. Secondary Outcome: Number of Participants With > 50% Lower Seizure Rate on PRX-0023.
Description: Participants used a seizure calendar to record the number of seizures that occurred during each three month treatment period, i.e., while participants were either on PRX-0023 or Placebo. Seizure rate was calculated as the total number of seizures occurring during the three month period. The number of participants with >50% lower seizure frequency during the active compared with the placebo period was determined.
Time Frame: Three months
Measure: Count of Participants; unit: Participants
Groups:
- All Participants Who Completed Study: All participants who completed both arms of the study
Arm/Group | All Participants Who Completed Study
Number analyzed (Participants) | 9
Participants | 0

3. Secondary Outcome: Mean Score on the Hamilton Anxiety Rating Scale at the End of the Active and Placebo Periods.
Description: Participants were administered the Hamilton Anxiety Rating Scale (HAM-A) at the end of each three month treatment period, i.e., while participants were either on PRX-0023 or Placebo. The HAM-A measures an individual's severity of anxiety symptoms. The scale consists of 14 parameters, each defined by a series of symptoms. Each group of symptoms is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where </=17 indicates mild anxiety, 18-24 mild to moderate anxiety and 25-30 moderate to severe anxiety and >30 severe anxiety.
Time Frame: Three months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PRX-0023 | Placebo
Number analyzed (Participants) | 9 | 10
score on a scale | 5.1 (5.0) | 5.7 (5.7)

4. Secondary Outcome: Mean Score on the Hamilton Depression Rating Scale at the End of the Active and Placebo Periods
Description: The Hamilton Depression Rating Scale (HAM-D) was administered to participants at the end of each treatment period. The HAM-D is a multiple item questionnaire used to provide an indication of depression. The questionnaire is designed for adults and is used to rate the severity of their depression by probing mood, feelings of guilt, suicide ideation, insomnia, agitation or retardation, anxiety, weight loss, and somatic symptoms. Although the HAM-D form lists 21 items, the scoring is based on the first 17 items. Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine items are scored from 0-2 with 0 = absent and 2 = frequent or severe. Scores range from 0 to 50 with a score of 0-7 representing normal and a score >/= 23 representing very severe depression.
Time Frame: Three months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PRX-0023 | Placebo
Number analyzed (Participants) | 9 | 10
score on a scale | 5.3 (3.9) | 8.6 (12.8)

5. Secondary Outcome: Mean Score on the Hopkins Verbal Learning Test-Revised (HVLT-R) at the End of the Active and Placebo Periods
Description: The HVLT-R is a word-list learning and memory test.The participant is read a list of words and asked to recall as many as possible, without regard to the order in which they were read.The list is read three times with recall requested after each presentation (immediate recall) and after a delay (delayed recall). Individual test results are compared to others of the same age (+/-5 years).Test results are presented as T-scores which are conventionally used in neuropsychology. The participant's raw scores are compared to a population expected raw score, for a particular age group. That score is converted to a T-score.The interpretation of these T-scores is such that 50 is representative of the normal score in that age group in the general population. The standard deviation of these distributions are 10 units. Therefore, a score between 30-40 is considered mildly impaired, 20-30 is indicative of severe problems with learning and memory and a score of 60-70 indicates a very good memory.
Time Frame: Three months
Population: Unable to complete the delayed recall in one participant in the placebo arm.
Measure: Mean (Standard Deviation); unit: psychometric T-score
Arm/Group | PRX-0023 | Placebo
Number analyzed (Participants) | 9 | 10
psychometric T-score
  Immediate Recall | 34.8 (13.8) | 41.6 (10.1)
  Delayed Recall: number analyzed (Participants) | 9 | 9
  Delayed Recall | 33.3 (14.1) | 39.2 (10.8)

6. Secondary Outcome: The Mean Score on the Brief Visuospatial Memory Test-Revised (BVMT-R), at the End of the Active and Placebo Period.
Description: The BVMT-R is a test of memory for visual information. Participants are shown a page with several geometric designs arranged in a 2x3 matrix and asked to study the designs. After the page is shown for a brief period the participant is asked to draw each figure.The same page is shown three times with recall requested after each presentation (immediate recall) and after a delay (delayed recall). Individual test results are compared to other people the same age (+/- 5 years).Test results are presented as T-scores which are conventionally used in neuropsychology. The participant's raw scores are compared to a population expected raw score, for a particular age group.That score is converted to a T-score.The interpretation of these T-scores is such that 50 is representative of the normal score in that age group in the general population.The standard deviation of these distributions are 10 units. A score of 30-40 is considered mildly impaired, 20-30 is indicative of severe problems
Time Frame: Three months
Population: Unable to complete the delayed recall in one subject in the placebo arm
Measure: Mean (Standard Deviation); unit: psychometric T-score
Arm/Group | PRX-0023 | Placebo
Number analyzed (Participants) | 9 | 10
psychometric T-score
  Immediate Recall | 37.4 (9.7) | 39.0 (9.9)
  Delayed Recall: number analyzed (Participants) | 9 | 9
  Delayed Recall | 38.0 (11.9) | 37.4 (15.4)

7. Secondary Outcome: Mean Score on the Columbia Suicide Severity Rating Scale at the End of the Active and Placebo Periods
Description: The Columbia Suicide Severity Rating Scale (C-SSRS) was administered to subjects at the end of each treatment period. The C-SSRS, is a suicidal ideation and behavior rating scale which evaluates suicide risk. The assessment rates an individual's degree of suicidal ideation on a scale, ranging from 0 to 6 as follows: 0 = No suicide ideation; 1 = Wish to be dead; 2 = Non-Specific Active Suicidal Thoughts; 3 = Active Suicidal Ideation with any methods (No Plan) without intent to act; 4 = Active Suicidal Ideation with some intent to act, without specific plan; 5 = Active Suicidal Ideation with specific plan and intent; and 6 = Actual Suicide Attempt
Time Frame: Three months
Population: Missing data for one participant in the Placebo group
Measure: Count of Participants; unit: Participants
Arm/Group | PRX-0023 | Placebo
Number analyzed (Participants) | 9 | 9
Participants
  0 | 9 | 8
  1 | 0 | 1
  2 | 0 | 0
  3 | 0 | 0
  4 | 0 | 0
  5 | 0 | 0
  6 | 0 | 0

8. Secondary Outcome: Results of Clinical Examination of the Nervous System at the End of the Active and Placebo Treatment Periods
Description: A clinical examination of the nervous system was administered by a physician to subjects at the end of each three month treatment period, i.e., while the participant was on PRX-0023 or Placebo. Results of the examination ranged from 0-4 with scores defined as follows: 0 = normal examination; 1 = Observation only; patient asymptomatic; 2 = Patient reports complaint associated with finding but no dysfunction; 3 = Patient reports some impairment of daily function associated with finding; 4 = Patient unable to carry out usual activities due to dysfunction associated with finding.
Time Frame: Three months
Measure: Count of Participants; unit: Participants
Groups:
- PRX-0023: Participants with epilepsy receiving PRX
Arm/Group | PRX-0023 | Placebo
Number analyzed (Participants) | 9 | 10
Participants
  0 | 8 | 9
  1 | 0 | 0
  2 | 1 | 1
  3 | 0 | 0
  4 | 0 | 0

9. Secondary Outcome: Results of Clinical Examination of the Respiratory System at the End of the Active and Placebo Treatment Periods
Description: A clinical examination of the respiratory system was administered by a physician to subjects at the end of each three month treatment period, i.e., while the participant was on PRX-0023 or Placebo. Results of the examination ranged from 0-4 with scores defined as follows: 0 = normal examination; 1 = Observation only; patient asymptomatic; 2 = Patient reports complaint associated with finding but no dysfunction; 3 = Patient reports some impairment of daily function associated with finding; 4 = Patient unable to carry out usual activities due to dysfunction associated with finding.
Time Frame: Three months
Measure: Count of Participants; unit: Participants
Arm/Group | PRX-0023 | Placebo
Number analyzed (Participants) | 9 | 10
Participants
  0 | 8 | 10
  1 | 1 | 0
  2 | 0 | 0
  3 | 0 | 0
  4 | 0 | 0

10. Secondary Outcome: Results of Clinical Examination of the Cardiovascular System at the End of the Active and Placebo Treatment Periods
Description: A clinical examination of the cardiovascular system was administered by a physician to subjects at the end of each three month treatment period, i.e., while the participant was on PRX-0023 or Placebo. Results of the examination ranged from 0-4 with scores defined as follows: 0 = normal examination; 1 = Observation only; patient asymptomatic; 2 = Patient reports complaint associated with finding but no dysfunction; 3 = Patient reports some impairment of daily function associated with finding; 4 = Patient unable to carry out usual activities due to dysfunction associated with finding.
Time Frame: Three months
Measure: Count of Participants; unit: Participants
Arm/Group | PRX-0023 | Placebo
Number analyzed (Participants) | 9 | 10
Participants
  0 | 8 | 9
  1 | 1 | 1
  2 | 0 | 0
  3 | 0 | 0
  4 | 0 | 0

11. Secondary Outcome: Results of Clinical Examination of the Musculoskeletal System at the End of the Active and Placebo Treatment Periods
Description: A clinical examination of the musculoskeletal system was administered by a physician to subjects at the end of each three month treatment period, i.e., while the participant was on PRX-0023 or Placebo. Results of the examination ranged from 0-4 with scores defined as follows: 0 = normal examination; 1 = Observation only; patient asymptomatic; 2 = Patient reports complaint associated with finding but no dysfunction; 3 = Patient reports some impairment of daily function associated with finding; 4 = Patient unable to carry out usual activities due to dysfunction associated with finding.
Time Frame: Three months
Measure: Count of Participants; unit: Participants
Arm/Group | PRX-0023 | Placebo
Number analyzed (Participants) | 9 | 10
Participants
  0 | 9 | 9
  1 | 0 | 1
  2 | 0 | 0
  3 | 0 | 0
  4 | 0 | 0

12. Secondary Outcome: Number of Subjects With an Abnormal CBC Result at the End of the Active and Placebo Periods
Description: A Complete Blood Count (CBC) was administered at the end of each three month treatment period. A complete blood count test measures several components and features of your blood, including: Red blood cells (which carry oxygen), White blood cells (which fight infection), Hemoglobin (the oxygen-carrying protein in red blood cells), Hematocrit (the proportion of red blood cells to the fluid component (plasma) in your blood), Platelets, (which help with blood clotting). Abnormal increases or decreases in cell counts as revealed in a complete blood count may indicate an underlying medical condition, i.e., anemia (abnormal red blood cells, hemoglobin, and/or hematocrit), leucopenia (a decrease in white blood cells), leucocytosis (an increase in white blood cells), and thrombocytosis (an increase in platelets). Results were classified as either normal or abnormal.
Time Frame: Three months
Measure: Count of Participants; unit: Participants
Arm/Group | PRX-0023 | Placebo
Number analyzed (Participants) | 9 | 10
Participants
  anemia | 2 | 1
  leucopenia | 2 | 1
  leucocytosis | 2 | 3
  thrombocytosis | 0 | 2

13. Secondary Outcome: Number of Subjects With Abnormal Clinical Chemistry Labs at the End of the Active and Placebo Periods
Description: The number of subjects with abnormal clinical chemistry labs which is defined as a value outside of the NIH Clinical Center normal range.
Time Frame: Three months
Measure: Count of Participants; unit: Participants
Arm/Group | PRX-0023 | Placebo
Number analyzed (Participants) | 9 | 10
Participants
  electrolyte abnormality | 4 | 4
  hyperglycemia | 2 | 1
  elevated liver function < 2 x normal | 3 | 3
  elevated liver function > 2 x normal | 1 | 0
  abnormal urinalysis | 3 | 4
  elevated uric acid | 0 | 1
  elevated BUN or Creatinine | 0 | 0

14. Secondary Outcome: Number of Subjects With an Abnormal ECG Result at the End of the Active and Placebo Periods
Description: An electrocardiogram was administered to participants at the end of each treatment period, i.e., at the end of the PRX-0023 and Placebo treatment periods. The number of abnormal ECG readings was noted in this measure.
Time Frame: Three months
Population: Missing data
Measure: Count of Participants; unit: Participants
Arm/Group | PRX-0023 | Placebo
Number analyzed (Participants) | 8 | 9
Participants | 2 | 3

ADVERSE EVENTS:
Time Frame: Adverse Events were collected following baseline history and physical examination and continued until study completion. Study duration was 42-46 weeks (+/- 4 weeks).
Arm/Group | PRX-0023 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 4/9 | 7/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRX-0023 (N=9) | Placebo (N=10)
Upper Respiratory Infection (Infections and infestations) | 2 (2) | 1 (1) — Chest cold, URI
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Small bumps on back (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Bumps at IV site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
GI Upset (Gastrointestinal disorders) | 1 (2) | 1 (1)
Gait Imbalance (Nervous system disorders) | 1 (1) | 0 (0)
Elevated liver function test >2x normal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Change in nails and hair (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Stomach flu (Infections and infestations) | 1 (1) | 0 (0)
Injury following seizure (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Bug bites (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 4 (4)
Weight gain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Increased appetite (Gastrointestinal disorders) | 0 (0) | 1 (2)
Achy and sweaty (Infections and infestations) | 0 (0) | 1 (1)
Chest pressure during sleep (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT01281956/Prot_SAP_000.pdf